CLINICAL TRIAL: NCT00325429
Title: A Multicenter, Open, Long Term Safety Study of 52 Weeks Treatment With Vildagliptin in Patients With Type 2 Diabetes
Brief Title: Long-Term Safety Study of Vildagliptin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A1304
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Vildagliptin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This study is not being conducted in the United States. Vildagliptin is an oral antidiabetic agent. This 52-week clinical study is designed as an open label, long-term study aimed to evaluate the safety of vildagliptin in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Patients who have been placed on diet and exercise therapy without achieving target blood glucose levels
* Outpatients

Exclusion Criteria:

* Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes
* Significant cardiovascular complications as defined by the protocol
* Significant diabetic complications as defined by the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-04

PRIMARY OUTCOMES:
Adverse events profile after 52 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline to endpoint on HbA1c at 52 weeks
Change from baseline to endpoint on fasting plasma glucose at 52 weeks
Change from baseline to endpoint in HOMA B at 52 weeks
Change from baseline to endpoint in HOMA IR at 52 weeks
Change from baseline to endpoint in body weight at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan